CLINICAL TRIAL: NCT04588415
Title: Supporting Family Members With Severe Grief Reaction During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Peter Lawlor, Clinician Investigator, Ottawa Hospital Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20200653-01H
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Bereavement; Severe Grief Reaction

STUDY DESIGN:
Intervention Model Description: All participants in the prospective bereavement data collection component of this study will be invited to participate in the virtual support group (VSG) intervention, regardless of the severity of their symptoms. Those with severe symptoms (indicated by an ICG-r score >25) will be notified that their symptoms are considered to be severe, with a suggestion to attend the VSGs. A recent meta-analysis of psychological interventions for grief found higher effect sizes in studies of participants who were >6 months post-loss, and those with higher baseline symptom levels. However, no participant in the study will be randomized to any treatment assignment, and the decision to attend the VSG will be left to the participants.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Support Group Arm (Experimental): Those with severe symptoms (indicated by an ICG-r score >25) will be notified that their symptoms are considered to be severe, with a suggestion to attend the virtual support groups. A recent meta-analysis of psychological interventions for grief found higher effect sizes in studies of participants who were >6 months post-loss, and those with higher baseline symptom levels. However, no participant in our study will be randomized to any treatment assignment, and the decision to attend the VSG will be left to the family members.
  Interventions: Other: Bereavement Virtual Support Group
- Non-Virtual Support Group Arm (No Intervention): Family members that choose not to participate in the Virtual Support Group will be part of this non-intervention arm

INTERVENTIONS:
Other: Bereavement Virtual Support Group — Family members who experience loss will be invited to attend a virtual support group (VSG) led by Bereaved Families of Ontario- Ottawa (BFO). In pre-COVID-19 times, BFO presented monthly "Support and Share" nights with guest speakers, followed by breakout peer support groups for all different types of losses: loss of child, spouse, parent, loss by suicide, etc. These groups are facilitated by trained volunteers with a shared loss and include between 75 and 150 participants. These Support and Share Nights serve as intake sessions- interested participants from the breakout groups can attend "Closed Groups" where a smaller group of participants (up to 12) explore their grief more deeply. These run over 8-10 consecutive weeks with the same group of participants. They are led by trained facilitators who have experienced similar losses. Each week has a different theme, based on evidence-based components of bereavement support (e.g. writing a letter to the deceased).
  Arms: Virtual Support Group Arm

SUMMARY:
This is a feasibility study taking place at The Ottawa Hospital (TOH), Hôpital Montfort, and Queensway Carleton Hospital that seeks to evaluate the impact of the COVID-19 pandemic on family member bereavement and study the effect of virtual support groups on reducing risk of developing Severe Grief Reaction (SGR). This project is inviting family members of deceased patients at either of the three before mentioned sites to enroll in this study.

DETAILED DESCRIPTION:
Background:

Severe grief reactions (SGR), or complicated grief (CG), are experienced by 2-3% of the population after the loss of a loved one, and can be associated with declining health, social distress, increased use of healthcare resources and higher mortality. SGR can be related to the circumstances of the patient at the end of life, particularly in deaths that were unexpected or traumatic, when the family member was unprepared or unsupported. The COVID-19 pandemic has affected many aspects of end-of-life care. For example, infection control measures may reduce interactions between long-term care residents and family members, and have often limited in-person family visiting to the final hours of life, or no visiting at all for patients with COVID-19. Anecdotally, this disruption of normal interactions has been difficult for patients and families alike, and it is known that isolation and lack of closure with a loved one can contribute to the risk of SGR. The prevalence of SGR is expected to rise amid increased challenges in supporting a surge of people with SGR due to physical distancing and limited bereavement resources.

Methods:

The proposed mixed methods explanatory study includes both retrospective and prospective data collection. The quantitative components will principally consist of natural experiments to identify patient/FM characteristics indicating a high risk of SGR during the COVID-19 pandemic. The qualitative components will deepen an understanding of the impact of COVID-19 on bereavement, while providing a formative evaluation for the virtual support groups. Study subjects will include all patients who died in an acute care facility in Ottawa (The Ottawa Hospital, Queensway-Carleton Hospital, and Hôpital Montfort) from January 1, 2020 until June 30, 2020, and their primary contact (as indicated in their medical record).

Significance:

Early identification of FMs at risk of SGR provides an opportunity for early intervention with the hope of preventing or reducing the severity of the SGR, but it also enables prioritization of those in greatest need, should demand exceed resources. Moreover, because it is still early in the pandemic, the study will be able to collect clinical data about the circumstances of the death, and consistently collect bereavement data for family members of people who died before and after the pandemic struck, and before and after the availability of virtual support groups. Therefore have a unique opportunity to conduct two natural experiments- studying the impact of the COVID pandemic on bereavement, and studying the effect of virtual support groups on symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Family Members of deceased patients from The Ottawa Hospital, Queensway-Carleton Hospital, and Hôpital Montfort

Exclusion Criteria:

* Anyone who is unable to participate in a virtual intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Downar, MD, Study Chair — Ottawa Hospital Research Institute; Peter G Lawlor, MD, Principal Investigator — Bruyere Continuing Care; Henrique Parsons, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified prior to entering analysis with anyone outside of the research team

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Support Group Arm: Those with severe symptoms (indicated by an ICG-r score >25) will be notified that their symptoms are considered to be severe, with a suggestion to attend the virtual support groups. A recent meta-analysis of psychological interventions for grief found higher effect sizes in studies of participants who were >6 months post-loss, and those with higher baseline symptom levels. No participant will be randomized to any treatment assignment. The decision to attend the VSG is left to the family members.
  Bereavement Virtual Support Group: Family members who experience loss will be invited to attend a virtual support group (VSG) led by Bereaved Families of Ontario- Ottawa (BFO). In pre-COVID-19 times, BFO presented monthly "Support and Share" nights with guest speakers, followed by breakout peer support groups for all different types of losses: loss of child, spouse, parent, loss by suicide, etc. These groups are facilitated by trained volunteers with a shared loss and include between 75 and 150 participants. These Support and Share Nights serve as intake sessions- participants from the breakout groups can attend "Closed Groups" where a smaller group of participants (up to 12) explore grief more deeply. These run over 8-10 consecutive weeks with the same group of participants. They are led by trained facilitators who have experienced similar losses. Each week has a different theme, based on evidence-based components of bereavement support (e.g. writing a letter to the deceased).
Period: Overall Study
Arm/Group | Virtual Support Group Arm | Non-Virtual Support Group Arm
Started | 0 | 121
Completed | 0 | 121
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants attended the virtual support group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Support Group Arm | Non-Virtual Support Group Arm | Total
Number analyzed (Participants) | 0 | 121 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 58.4 (14.7) | 58.4 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 80 | 80
  Male |  | 41 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian |  | 92 | 92
  Asian |  | 13 | 13
  African, Caribbean, or non-specified Black |  | 7 | 7
  Latin, Central, and South American |  | 4 | 4
  Indigenous (First Nations, Métis, non-status) |  | 3 | 3
  Mixed (Jamaican and French, German and Jamaican) |  | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada |  | 121 | 121
Physical presence of family in the last 48 h of life [Count of Participants; unit: Participants]
  Yes |  | 95 | 95
  No |  | 26 | 26
Virtual presence of family in the last 48 h of life [Count of Participants; unit: Participants]
  Yes |  | 18 | 18
  No |  | 103 | 103
Physical/in person interaction between the team and family in the last 5 days of life [Mean (Standard Deviation); unit: Number of interactions] — Total number of physical/in-person interactions between the healthcare team and decedents' family members in the last 5 days of life
  Number of interactions |  | 3 (3.3) | 3 (3.3)
Brief Family Relationship Scale (Total score) [Mean (Standard Deviation); unit: units on a scale] — A 16-item measure with each item rated as a yes or no (1 or 0). Higher total scores indicate higher levels of family functioning. Total scores range from 0-16.
  units on a scale |  | 14.0 (2.2) | 14.0 (2.2)
Relationship to deceased [Count of Participants; unit: Participants]
  Spouse/partner |  | 24 | 24
  Child |  | 75 | 75
  Sibling |  | 9 | 9
  Friend |  | 2 | 2
  Other |  | 11 | 11
Phone call interaction between the team and family in the last 5 days of life [Mean (Standard Deviation); unit: Number of interactions] — Total number of phone call interactions between the healthcare team and decedents' family members in the last 5 days of life
  Number of interactions |  | 2.3 (2.4) | 2.3 (2.4)
Virtual interaction between the team and family in the last 5 days of life [Mean (Standard Deviation); unit: Number of interactions] — Total number of virtual interactions between the healthcare team and decedents' family members in the last 5 days of life
  Number of interactions |  | 0.2 (0.7) | 0.2 (0.7)
ICU admission [Count of Participants; unit: Participants]
  Yes |  | 39 | 39
  No |  | 82 | 82
Intubation [Count of Participants; unit: Participants]
  Yes |  | 25 | 25
  No |  | 96 | 96
Decedent age [Mean (Standard Deviation); unit: years] |  | 80.1 (13.1) | 80.1 (13.1)
Decedent sex [Count of Participants; unit: Participants]
  Male |  | 67 | 67
  Female |  | 54 | 54
Death disposition [Count of Participants; unit: Participants]
  Medicine |  | 88 | 88
  ICU |  | 33 | 33
Days in hospital [Mean (Standard Deviation); unit: days] |  | 12.0 (18.0) | 12.0 (18.0)
Participant education [Count of Participants; unit: Participants]
  Did not complete high school |  | 1 | 1
  High school (some or all) |  | 26 | 26
  Post-secondary education |  | 94 | 94
Participant marital status [Count of Participants; unit: Participants]
  Single |  | 20 | 20
  Common-law |  | 11 | 11
  Married |  | 53 | 53
  Separated |  | 4 | 4
  Divorced |  | 8 | 8
  Widowed |  | 25 | 25

OUTCOME MEASURES:

1. Primary Outcome: The Inventory for Complicated Grief-revised (ICG-r) Score at 6 Months Post-death
Description: This tool, used to detect pathological grief, has a total of 19 questions. Respondents rate the frequency with which they experience each item on a 5-point scale (0-4), ranging from "never" to "always." Respondents with ICG-r scores greater than 25 are significantly more impaired in social, general, mental and physical health functioning and in bodily pain than those with ICG-r scores less than or equal to 25. Higher scores result in higher likelihood of CG.
Time Frame: at 6 months post-death
Population: No participants indicated they attended a virtual support group.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Support Group Arm | Non-Virtual Support Group Arm
Number analyzed (Participants) | 0 | 121
Participants
  ICG total score >25 |  | 35
  ICG total score ≤ 25 |  | 86

2. Primary Outcome: The Inventory for Complicated Grief-revised (ICG-r) Score at 12 Months Post-death
Description: Participating FMs will have a repeat ICG-r assessment (as described for primary outcome #1) at 12 months post-death.
Time Frame: at 12 months post-death
Population: No participants indicated they attended a virtual support group. Of the 121 participants who completed the baseline grief assessment, 111 completed the follow-up assessment at 12-months post death.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Support Group Arm | Non-Virtual Support Group Arm
Number analyzed (Participants) | 0 | 111
Participants
  ICG >25 at follow-up |  | 32
  ICG ≤25 at follow-up |  | 79

3. Primary Outcome: Change in ICG-r Score From 6 Months to 12 Months Post-death
Description: The relative changes in ICG-r scores (change in mean score with SD) between 6 and 12 months of family members who participate in the VSGs vs. those who do not will be compared as a measure of the efficacy of the VSG intervention
Time Frame: at 12 months post-death relative to 6 months post-death
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Support Group Arm | Non-Virtual Support Group Arm
Number analyzed (Participants) | 0 | 111
score on a scale |  | -0.01 (8.5)

4. Primary Outcome: Qualitative Interviews Post-Virtual Support Group
Description: The data for this primary outcome could not be collected due to no participants completing the virtual support group intervention. As a result, no interviews could be conducted. Interviews with family member participants upon completion of the virtual support group intervention were to be conducted to determine usefulness for family members' bereavement process. This is a qualitative method of data collection so there is no scale or score.
Time Frame: Through study completion, an average of 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 12 months post-death
Description: No adverse events were reported
Arm/Group | Virtual Support Group Arm | Non-Virtual Support Group Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/121
Other Adverse Events (participants affected / at risk) | 0/0 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT04588415/Prot_SAP_000.pdf